CLINICAL TRIAL: NCT01004861
Title: A Phase 1 Study to Assess Safety, Pharmacokinetics, and Pharmacodynamics of PLX3397 in Patients With Advanced, Incurable, Solid Tumors in Which the Target Kinases Are Linked to Disease Pathophysiology
Brief Title: Safety Study of PLX108-01 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Plexxikon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLX108-01
Record Dates: First submitted 2009-10-28; First posted 2009-10-30 (Estimated); Results first posted 2020-04-06 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Solid Tumor
Keywords: PVNS
MeSH Terms: interventions — pexidartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PLX3397 (Experimental)
  Interventions: Drug: PLX3397

INTERVENTIONS:
Drug: PLX3397 — Capsules administered once or twice daily, continuous dosing

SUMMARY:
PLX3397 is a selective inhibitor of Fms, Kit, and oncogenic Flt3 activity. The primary objective of this study is to evaluate the safety and pharmacokinetics of orally administered PLX3397 in patients with advanced, incurable, solid tumors in which these target kinases are linked to disease pathophysiology. The secondary objective is to measure the pharmacodynamic activity of PLX3397 via blood, plasma and urine biomarkers of Fms activity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Solid tumors refractory to standard therapy
* For the Extension cohorts, patients must have measurable disease by RECIST criteria and meet the following disease-specific criteria:

  * For advanced or recurrent mucoepidermal carcinoma (MEC) of the salivary gland, patients must not be candidates for curative surgery or radiotherapy.
  * For pigmented villo-nodular synovitis (PVNS), patients must have a histologically confirmed diagnosis of inoperable progressive or relapsing PVNS, or resectable tumor requesting mutilating surgery, as well as demonstrated progressive disease in the last 12 months.
  * For gastrointestinal stromal tumors (GIST), patients must have failed previous therapy with imatinib and sunitinib. Patients with known PDGFR mutations are excluded, but mutation testing is not required for study entry.
  * For anaplastic thyroid cancer (ATC), patients must have histologically or cytologically diagnosed advanced ATC.
  * For metastatic solid tumors with documented malignant pleural and/or peritoneal effusions, patients must not be receiving specific therapy for the effusion or have an indwelling drain.
* Eastern Cooperative Oncology Group performance status 0 or 1
* Life expectancy >= 3 months
* Adequate hepatic, renal, and bone marrow function

Exclusion Criteria:

* Specific anti-cancer therapy within 3 weeks of study start
* Uncontrolled intercurrent illness
* Refractory nausea or vomiting, or malabsorption
* Mean corrected QT interval (QTc) >= 450 msec (for males) or QTc >= 470 msec (for females)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2009-10-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Daiichi Sankyo
Locations (13):
- United States (13):
  - HonorHealth, Scottsdale, Arizona
  - UCLA, Los Angeles, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Memorial Sloan-Kettering Cancer Center (MSKCC), New York, New York
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Medical Center, Nashville, Tennessee
  - Texas Oncology, PA (North), Dallas, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Evergreen Hematology & Oncology, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Tap WD, Singh AS, Anthony SP, Sterba M, Zhang C, Healey JH, Chmielowski B, Cohn AL, Shapiro GI, Keedy VL, Wainberg ZA, Puzanov I, Cote GM, Wagner AJ, Braiteh F, Sherman E, Hsu HH, Peterfy C, Gelhorn HL, Ye X, Severson P, West BL, Lin PS, Tong-Starksen S. Results from Phase I Extension Study Assessing Pexidartinib Treatment in Six Cohorts with Solid Tumors including TGCT, and Abnormal CSF1 Transcripts in TGCT. Clin Cancer Res. 2022 Jan 15;28(2):298-307. doi: 10.1158/1078-0432.CCR-21-2007. Epub 2021 Oct 29. PMID 34716196
- [Derived] Lewis JH, Gelderblom H, van de Sande M, Stacchiotti S, Healey JH, Tap WD, Wagner AJ, Pousa AL, Druta M, Lin CC, Baba HA, Choi Y, Wang Q, Shuster DE, Bauer S. Pexidartinib Long-Term Hepatic Safety Profile in Patients with Tenosynovial Giant Cell Tumors. Oncologist. 2021 May;26(5):e863-e873. doi: 10.1002/onco.13629. Epub 2020 Dec 24. PMID 33289960
- [Derived] Tap WD, Wainberg ZA, Anthony SP, Ibrahim PN, Zhang C, Healey JH, Chmielowski B, Staddon AP, Cohn AL, Shapiro GI, Keedy VL, Singh AS, Puzanov I, Kwak EL, Wagner AJ, Von Hoff DD, Weiss GJ, Ramanathan RK, Zhang J, Habets G, Zhang Y, Burton EA, Visor G, Sanftner L, Severson P, Nguyen H, Kim MJ, Marimuthu A, Tsang G, Shellooe R, Gee C, West BL, Hirth P, Nolop K, van de Rijn M, Hsu HH, Peterfy C, Lin PS, Tong-Starksen S, Bollag G. Structure-Guided Blockade of CSF1R Kinase in Tenosynovial Giant-Cell Tumor. N Engl J Med. 2015 Jul 30;373(5):428-37. doi: 10.1056/NEJMoa1411366. PMID 26222558

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The dose escalation phase administered ascending daily oral doses of PLX3397 to patients with solid tumors and evaluated PK and toxicity. Once the recommended phase 2 dose was reached, 6 extension cohorts were enrolled, consisting of a variety of tumor types.
Pre-assignment Details: At least 3 participants and up to 6 participants were to be enrolled in each dose level using 100% dose increments for each level in the absence of Grade 2 or greater drug-attributable toxicity. Dose escalation was only permitted if adequate safety and tolerability were observed at the previous lower dose for 28 days for the first 3 participants.
Groups:
- Dose Escalation Cohort 1: 200 mg QD: Participants with advanced, incurable, solid tumors who received PLX3397 200 mg QD.
- Dose Escalation Cohort 2: 300 mg QD: Participants with advanced, incurable, solid tumors who received PLX3397 300 mg QD.
- Dose Escalation Cohort 3: 400 mg QD: Participants with advanced, incurable, solid tumors who received PLX3397 400 mg QD.
- Dose Escalation Cohort 4: 600 mg QD: Participants with advanced, incurable, solid tumors who received PLX3397 600 mg QD.
- Dose Escalation Cohort 5: 900 mg/Day (500mg AM, 400mg PM): Participants with advanced, incurable, solid tumors who received PLX3397 900 mg/day.
- Dose Escalation Cohort 6: 1200 mg/Day (600mg BID): Participants with advanced, incurable, solid tumors who received PLX3397 1200 mg/day.
- Dose Escalation Cohort 7: 1000 mg/Day (500mg BID): Participants with advanced, incurable, solid tumors who received PLX3397 1000 mg/day.
- Dose Extension: MEC Cohort 1000 mg/Day (600mg AM, 400mg PM): Participants with advanced or recurrent mucoepidermoid carcinoma (MEC) who received PLX3397.
- Dose Extension: PVNS Cohort PVNS Cohort 1000 mg/Day (600mg AM, 400mg PM): Participants with advanced pigmented villonodular synovitis (PVNS) who received PLX3397.
- Dose Extension: GIST Cohort 1000 mg/Day (600mg AM, 400mg PM): Participants with advanced gastrointestinal stromal tumor (GIST) who received PLX3397.
- Dose Extension: ATC Cohort 1000 mg/Day (600mg AM, 400mg PM): Participants with anaplastic thyroid carcinoma (ATC) who received PLX3397.
- Dose Extension: Malignant Effusion Cohort 1000 mg/Day (600mg AM, 400mg PM): Participants with advanced solid tumors with malignant effusion who received PLX3397.
- Dose Extension: Other Tumors 1000 mg/Day (600mg AM, 400mg PM): Participants with other solid tumor types who received PLX3397.
Period: Overall Study
Arm/Group | Dose Escalation Cohort 1: 200 mg QD | Dose Escalation Cohort 2: 300 mg QD | Dose Escalation Cohort 3: 400 mg QD | Dose Escalation Cohort 4: 600 mg QD | Dose Escalation Cohort 5: 900 mg/Day (500mg AM, 400mg PM) | Dose Escalation Cohort 6: 1200 mg/Day (600mg BID) | Dose Escalation Cohort 7: 1000 mg/Day (500mg BID) | Dose Extension: MEC Cohort 1000 mg/Day (600mg AM, 400mg PM) | Dose Extension: PVNS Cohort PVNS Cohort 1000 mg/Day (600mg AM, 400mg PM) | Dose Extension: GIST Cohort 1000 mg/Day (600mg AM, 400mg PM) | Dose Extension: ATC Cohort 1000 mg/Day (600mg AM, 400mg PM) | Dose Extension: Malignant Effusion Cohort 1000 mg/Day (600mg AM, 400mg PM) | Dose Extension: Other Tumors 1000 mg/Day (600mg AM, 400mg PM)
Started | 3 | 6 | 6 | 6 | 7 | 6 | 7 | 4 | 39 | 11 | 9 | 8 | 20
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 6 | 6 | 7 | 6 | 7 | 4 | 39 | 11 | 9 | 8 | 20
Not completed — Disease progression | 3 | 4 | 5 | 4 | 4 | 4 | 5 | 1 | 4 | 7 | 6 | 3 | 8
Not completed — Physician Decision | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 13 | 1 | 1 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0
Not completed — Non-compliance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 3
Not completed — Patient decision | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 7 | 1 | 1 | 2 | 3
Not completed — Transitioned to Phase 4 study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Patient completed 12-week follow-up and continued on commercially approved drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Patient withdrew | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Surgical resection | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Patient maintained complete response status throughout drug holiday | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Study termination by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Escalation Cohort 5: 900 mg/Day: Participants with advanced, incurable, solid tumors who received PLX3397 900 mg/day.
- Dose Escalation Cohort 6: 1200 mg/Day: Participants with advanced, incurable, solid tumors who received PLX3397 1200 mg/day.
- Dose Escalation Cohort 7: 1000 mg/Day: Participants with advanced, incurable, solid tumors who received PLX3397 1000 mg/day.
- Dose Extension: MEC Cohort: Participants with advanced mucoepidermoid carcinoma (MEC) who received PLX3397.
- Dose Extension: PVNS Cohort: Participants with advanced pigmented villonodular synovitis (PVNS) who received PLX3397.
- Dose Extension: GIST Cohort: Participants with advanced gastrointestinal stromal tumor (GIS) who received PLX3397.
- Dose Extension: ATC Cohort: Participants with anaplastic thyroid carcinoma (ATC) who received PLX3397.
- Dose Extension: Malignant Effusion Cohort: Participants with advanced solid tumors with malignant effusion who received PLX3397.
- Dose Extension: Other Solid Tumor Type Cohort: Participants with other solid tumor types who received PLX3397.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Cohort 1: 200 mg QD | Dose Escalation Cohort 2: 300 mg QD | Dose Escalation Cohort 3: 400 mg QD | Dose Escalation Cohort 4: 600 mg QD | Dose Escalation Cohort 5: 900 mg/Day | Dose Escalation Cohort 6: 1200 mg/Day | Dose Escalation Cohort 7: 1000 mg/Day | Dose Extension: MEC Cohort | Dose Extension: PVNS Cohort | Dose Extension: GIST Cohort | Dose Extension: ATC Cohort | Dose Extension: Malignant Effusion Cohort | Dose Extension: Other Solid Tumor Type Cohort | Total
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 7 | 6 | 7 | 4 | 39 | 11 | 9 | 8 | 20 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 2 | 3 | 5 | 3 | 5 | 4 | 37 | 8 | 3 | 4 | 15 | 93
  >=65 years | 1 | 4 | 4 | 3 | 2 | 3 | 2 | 0 | 2 | 3 | 6 | 4 | 5 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (10.1) | 65.7 (2.3) | 63.5 (8.6) | 61.5 (19.1) | 52.3 (15.0) | 56.3 (17.1) | 50.4 (19.8) | 47.3 (18.4) | 45.1 (14.0) | 57.6 (12.1) | 65.9 (14.7) | 58.1 (13.3) | 52.0 (15.1) | 58.3 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 3 | 3 | 4 | 3 | 6 | 1 | 22 | 6 | 4 | 5 | 5 | 68
  Male | 1 | 2 | 3 | 3 | 3 | 3 | 1 | 3 | 17 | 5 | 5 | 3 | 15 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 5
  White | 3 | 6 | 6 | 6 | 7 | 5 | 7 | 4 | 33 | 10 | 8 | 8 | 18 | 121
  Black of African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Multiple races | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 6 | 6 | 7 | 6 | 7 | 4 | 39 | 11 | 9 | 8 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Summary of Derived Best Tumor Response Per the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 - Dose Escalation (Efficacy Evaluable Population)
Description: Best overall tumor response (complete response [CR], partial response [PR], stable disease [SD], progressive disease [PD]) is reported, including participants who were not evaluable (NE).
  RECIST v1.1 for target lesions are assessed by magnetic resonance imaging, computed tomography, or positron emission tomography-computed tomography and are summarized as: CR, Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm; PR, At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; PD, at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (includes the baseline sum). In addition, the sum must also demonstrate an absolute increase of at least 5 mm; SD, Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Every 2 months beginning Cycle 3, Day 1 until disease progression (up to approximately 30 months postdose)
Population: Best overall tumor response was assessed in the Efficacy Evaluable Population.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All participants with advanced, incurable, solid tumors who received PL3397.
Arm/Group | Dose Escalation Cohort 1: 200 mg QD | Dose Escalation Cohort 2: 300 mg QD | Dose Escalation Cohort 3: 400 mg QD | Dose Escalation Cohort 4: 600 mg QD | Dose Escalation Cohort 5: 900 mg/Day (500mg AM, 400mg PM) | Dose Escalation Cohort 6: 1200 mg/Day (600mg BID) | Dose Escalation Cohort 7: 1000 mg/Day (500mg BID) | All Participants
Number analyzed (Participants) | 3 | 5 | 5 | 5 | 6 | 5 | 6 | 35
Participants
  Censored participants | 0 | 1 | 2 | 0 | 3 | 0 | 3 | 9
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  SD | 0 | 1 | 0 | 2 | 3 | 1 | 1 | 8
  PD | 3 | 4 | 3 | 3 | 2 | 4 | 3 | 22
  NE | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 4

2. Primary Outcome: Summary of Derived Best Tumor Response Per the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 - Dose Extension (Efficacy Evaluable Population)
Description: as for outcome 1
Time Frame: Every 2 months beginning Cycle 3, Day 1 until disease progression (up to approximately 30 months postdose)
Population: Best overall tumor response was assessed in the Efficacy Evaluable Population.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Extension: GIST Cohort: Participants with advanced gastrointestinal stromal tumor (GIST) who received PLX3397.
Arm/Group | Dose Extension: MEC Cohort | Dose Extension: PVNS Cohort | Dose Extension: GIST Cohort | Dose Extension: ATC Cohort | Dose Extension: Malignant Effusion Cohort | Dose Extension: Other Solid Tumor Type Cohort
Number analyzed (Participants) | 2 | 37 | 9 | 6 | 6 | 14
Participants
  CR | 0 | 2 | 0 | 0 | 0 | 0
  PR | 0 | 22 | 0 | 0 | 0 | 1
  SD | 1 | 8 | 4 | 0 | 3 | 7
  PD | 1 | 1 | 5 | 6 | 2 | 6
  NE | 0 | 4 | 0 | 0 | 1 | 0
  Overall response rate (CR or PR) | 0 | 24 | 0 | 0 | 0 | 1

3. Primary Outcome: Duration of Response (Efficacy Evaluable Population) - Dose Extension
Description: Duration of Response (DOR) is defined as the number of days from the date of initial response (CR or PR confirmed at least 28 days later) to the date of first documented disease progression/relapse or death, whichever occurs first. If no disease progression or death is documented prior to study termination, analysis cutoff, or the start of confounding anticancer therapy, DOR is censored as of the date of their last imaging exam of target or non-target lesions prior to post-surgery and/or off-treatment scans.
Time Frame: From initial response until disease progression or death, up to approximately 30 months postdose
Population: Duration of response was assessed among participants with response of CR or PR in the Efficacy Evaluable Population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dose Extension: MEC Cohort | Dose Extension: PVNS Cohort | Dose Extension: GIST Cohort | Dose Extension: ATC Cohort | Dose Extension: Malignant Effusion Cohort | Dose Extension: Other Solid Tumor Type Cohort
Number analyzed (Participants) | 0 | 24 | 0 | 0 | 0 | 1
days |  | NA [943 to NA] — Lack of median value is due to <50% of the participants experiencing the event. In a Kaplan-Meier analysis, the curve would never fall below the 50% mark, and would continue to the largest observed censored time value. |  |  |  | 115 [NA to NA] — There were not enough events to estimate a 95% confidence interval for the median survival time.

4. Primary Outcome: Progression-free Survival (Efficacy Evaluable Population) - Dose Extension
Description: Progression-Free Survival (PFS) is defined as the number of days from the first day of treatment to the first documented disease progression or date of death, whichever occurs first. If no disease progression or death is documented prior to study termination, analysis cutoff, or the start of confounding anticancer therapy, PFS is censored at the date of last evaluable tumor assessment.
Time Frame: From Cycle 1 Day 1 to disease progression or death
Population: Progression-free survival was assessed in the Efficacy Evaluable Population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dose Extension: MEC Cohort | Dose Extension: PVNS Cohort | Dose Extension: GIST Cohort | Dose Extension: ATC Cohort | Dose Extension: Malignant Effusion Cohort | Dose Extension: Other Solid Tumor Type Cohort
Number analyzed (Participants) | 2 | 37 | 9 | 6 | 6 | 14
days | NA [43 to NA] — Insufficient number of events; Lack of median value is due to 50% or fewer participants experiencing the event. In a Kaplan-Meier analysis, the curve would never fall below the 50% mark, and would continue to the largest observed censored time value. | NA [667 to NA] — Insufficient number of events; Lack of median value is due to 50% or fewer participants experiencing the event. In a Kaplan-Meier analysis, the curve would never fall below the 50% mark, and would continue to the largest observed censored time value. | 54 [40 to 164] | 50 [34 to 56] | 78 [51 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it is NA. | 161 [54 to 504]

5. Primary Outcome: Best Overall Tumor Response (PVNS Cohort) Per the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 - Dose Extension
Description: as for outcome 1
Time Frame: Every 2 months beginning Cycle 3, Day 1 until disease progression
Population: Best overall tumor response was assessed in the Efficacy Evaluable Population.
Measure: Count of Participants; unit: Participants
Groups:
- PVNS Cohort: Participants with advanced pigmented villonodular synovitis (PVNS) who received PLX3397.
Arm/Group | PVNS Cohort
Number analyzed (Participants) | 37
Participants
  CR | 2
  PR | 22
  SD | 8
  PD | 1
  NE | 4
  Overall response rate (CR or PR) | 24

6. Primary Outcome: Summary Statistics for Selected PLX3397 Pharmacokinetics Parameter Cmax, Study Day Cycle 1 Day 15, Stratified by Cohort - Dose Escalation
Description: Cycle 1 Day 15 pharmacokinetic (PK) timepoints taken are: For once daily (QD) dosing, obtained predose (morning) and 0.5, 1, 2, 4, and 8 hours postdose. For twice a day (BID) dosing predose (morning) and 1, 2, 4, and 7 hours postdose. The second dose will then be administered, and PK obtained 1 hour post the second dose (8 hours post the first dose). For BID dosing, no run-in is planned.
Time Frame: Cycle 1, Day 15
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Dose Escalation Cohort 1: 200 mg QD | Dose Escalation Cohort 2: 300 mg QD | Dose Escalation Cohort 3: 400 mg QD | Dose Escalation Cohort 4: 600 mg QD | Dose Escalation Cohort 5: 900 mg/Day (500mg AM, 400mg PM) | Dose Escalation Cohort 6: 1200 mg/Day (600mg BID) | Dose Escalation Cohort 7: 1000 mg/Day (500mg BID)
Number analyzed (Participants) | 3 | 5 | 5 | 5 | 6 | 5 | 6
ng/mL | 1730 [1460 to 2900] | 3630 [1360 to 5300] | 3160 [2140 to 5210] | 6570 [4000 to 14300] | 6290 [5520 to 10400] | 10600 [5070 to 12500] | 6320 [5920 to 10100]

7. Primary Outcome: Summary Statistics for Selected PLX3397 Pharmacokinetics Parameter Tmax, Study Day Cycle 1 Day 15, Stratified by Cohort - Dose Escalation
Description: Cycle 1 Day 15 PK timepoints taken are: For QD dosing, obtained predose (morning) and 0.5, 1, 2, 4, and 8 hours postdose. For BID dosing predose (morning) and 1, 2, 4, and 7 hours postdose. The second dose will then be administered, and PK obtained 1 hour post the second dose (8 hours post the first dose). For BID dosing, no run-in is planned.
Time Frame: Cycle 1, Day 15
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hour
Arm/Group | Dose Escalation Cohort 1: 200 mg QD | Dose Escalation Cohort 2: 300 mg QD | Dose Escalation Cohort 3: 400 mg QD | Dose Escalation Cohort 4: 600 mg QD | Dose Escalation Cohort 5: 900 mg/Day (500mg AM, 400mg PM) | Dose Escalation Cohort 6: 1200 mg/Day (600mg BID) | Dose Escalation Cohort 7: 1000 mg/Day (500mg BID)
Number analyzed (Participants) | 3 | 5 | 5 | 5 | 6 | 5 | 6
hour | 2.00 [1.08 to 4.00] | 1.97 [0.58 to 2.03] | 0.98 [0.50 to 2.20] | 1.04 [0.50 to 2.03] | 2.00 [0 to 2.03] | 1.05 [1.00 to 4.17] | 2.03 [0 to 6.95]

8. Primary Outcome: Summary Statistics for Selected PLX3397 Pharmacokinetics Parameter Area Under the Curve (AUC0-24), Study Day Cycle 1 Day 15, Stratified by Cohort - Dose Escalation
Description: Cycle 1 Day 15 PK timepoints taken are: For QD dosing, obtained predose (morning) and 0.5, 1, 2, 4, and 8 hours postdose. For BID dosing, predose (morning) and 1, 2, 4, and 7 hours postdose. The second dose will then be administered, and PK obtained 1 hour post the second dose (8 hours post the first dose). For BID dosing, no run-in is planned.
Time Frame: Cycle 1, Day 15 (QD dosing: predose [morning] and 0.5, 1, 2, 4, and 8 hours postdose; BID dosing: predose [morning] and 1, 2, 4, and 7 hours postdose)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: ng*hr/mL
Arm/Group | Dose Escalation Cohort 1: 200 mg QD | Dose Escalation Cohort 2: 300 mg QD | Dose Escalation Cohort 3: 400 mg QD | Dose Escalation Cohort 4: 600 mg QD | Dose Escalation Cohort 5: 900 mg/Day (500mg AM, 400mg PM) | Dose Escalation Cohort 6: 1200 mg/Day (600mg BID) | Dose Escalation Cohort 7: 1000 mg/Day (500mg BID)
Number analyzed (Participants) | 3 | 5 | 5 | 5 | 6 | 5 | 6
ng*hr/mL | 26200 [13200 to 37100] | 50400 [19500 to 83100] | 40500 [29500 to 57300] | 81000 [74300 to 166000] | 107000 [68400 to 139000] | 173000 [80200 to 190000] | 115000 [105000 to 226000]

9. Primary Outcome: Numeric Rating Scale (NRS) for PVNS Symptoms Sum of Scores Through Cycle 2 (Efficacy Evaluable Population) - Dose Extension
Description: The NRS for PVNS Symptoms instrument is a 5-item self-administered questionnaire to assess the "worst" of each of the symptoms pain, swelling, stiffness, instability and limited motion in the last 24 hours. A 0 to 10 NRS is provided for each symptom. For pain, 0 indicates "no pain" and 10 indicates "pain as bad as you can imagine". For the other 4 symptoms, 0 indicates "no (symptom)" and 10 indicates "(symptom) worst imaginable", e.g., "swelling - worst imaginable." Higher scores indicated worse outcome.
Time Frame: Baseline, Cycle 1 Day 15, Cycle 2, Cycle 3, Cycle 12, Cycle 24, Cycle 36, and Cycle 46 (each cycle was 28 days)
Population: NRS for PVNS symptoms were assessed in patients with available data in the Efficacy Evaluable Population.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- NRS for PVNS Symptoms Evaluable Population: Participants who were administered the NRS scale at baseline and monthly on treatment.
Arm/Group | NRS for PVNS Symptoms Evaluable Population
Number analyzed (Participants) | 21
units on a scale
  Pain; Baseline | 5.2 (2.1)
  Pain; Cycle 1 Day 15 | 3.5 (2.9)
  Pain; Cycle 2 | 3.6 (2.6)
  Pain; Cycle 3: number analyzed (Participants) | 20
  Pain; Cycle 3 | 2.3 (1.9)
  Pain; Cycle 12: number analyzed (Participants) | 15
  Pain; Cycle 12 | 1.3 (1.8)
  Pain; Cycle 24: number analyzed (Participants) | 11
  Pain; Cycle 24 | 1.5 (1.4)
  Pain; Cycle 36: number analyzed (Participants) | 9
  Pain; Cycle 36 | 2.0 (2.8)
  Pain; Cycle 46: number analyzed (Participants) | 8
  Pain; Cycle 46 | 1.8 (2.0)
  Swelling; Baseline | 4.7 (2.9)
  Swelling; Cycle 1 Day 15 | 3.1 (2.5)
  Swelling; Cycle 2 | 2.6 (2.3)
  Swelling; Cycle 3: number analyzed (Participants) | 20
  Swelling; Cycle 3 | 1.5 (1.4)
  Swelling; Cycle 12: number analyzed (Participants) | 15
  Swelling; Cycle 12 | 0.8 (1.2)
  Swelling; Cycle 24: number analyzed (Participants) | 11
  Swelling; Cycle 24 | 0.8 (0.8)
  Swelling; Cycle 36: number analyzed (Participants) | 9
  Swelling; Cycle 36 | 1.2 (1.8)
  Swelling; Cycle 46: number analyzed (Participants) | 8
  Swelling; Cycle 46 | 1.1 (1.2)
  Stiffness; Baseline | 4.7 (2.9)
  Stiffness; Cycle 1 Day 15 | 3.6 (2.9)
  Stiffness; Cycle 2 | 3.1 (2.7)
  Stiffness; Cycle 3: number analyzed (Participants) | 20
  Stiffness; Cycle 3 | 2.2 (1.9)
  Stiffness; Cycle 12: number analyzed (Participants) | 15
  Stiffness; Cycle 12 | 1.5 (1.9)
  Stiffness; Cycle 24: number analyzed (Participants) | 11
  Stiffness; Cycle 24 | 1.2 (1.1)
  Stiffness; Cycle 36: number analyzed (Participants) | 9
  Stiffness; Cycle 36 | 1.6 (2.1)
  Stiffness; Cycle 46: number analyzed (Participants) | 8
  Stiffness; Cycle 46 | 1.6 (1.6)
  Instability; Baseline | 2.9 (2.6)
  Instability; Cycle 1 Day 15 | 2.1 (2.6)
  Instability; Cycle 2 | 2.1 (2.5)
  Instability; Cycle 3: number analyzed (Participants) | 20
  Instability; Cycle 3 | 1.2 (1.4)
  Instability; Cycle 12: number analyzed (Participants) | 15
  Instability; Cycle 12 | 0.8 (1.0)
  Instability; Cycle 24: number analyzed (Participants) | 11
  Instability; Cycle 24 | 0.4 (0.7)
  Instability; Cycle 36: number analyzed (Participants) | 9
  Instability; Cycle 36 | 0.4 (0.7)
  Instability; Cycle 46: number analyzed (Participants) | 8
  Instability; Cycle 46 | 0.4 (0.7)
  Limited motion; Baseline | 4.8 (2.8)
  Limited motion; Cycle 1 Day 15 | 3.2 (2.7)
  Limited motion; Cycle 2 | 3.0 (2.4)
  Limited motion; Cycle 3: number analyzed (Participants) | 20
  Limited motion; Cycle 3 | 1.9 (1.7)
  Limited motion; Cycle 12: number analyzed (Participants) | 15
  Limited motion; Cycle 12 | 1.4 (1.7)
  Limited motion; Cycle 24: number analyzed (Participants) | 11
  Limited motion; Cycle 24 | 1.0 (1.0)
  Limited motion; Cycle 36: number analyzed (Participants) | 9
  Limited motion; Cycle 36 | 1.7 (2.3)
  Limited Motion; Cycle 46: number analyzed (Participants) | 8
  Limited Motion; Cycle 46 | 1.8 (1.7)

ADVERSE EVENTS:
Time Frame: Adverse events (and serious adverse events) were recorded from the time the participant received the first dose of study drug up to 30 days after the last dose, up to approximately 30 months postdose.
Groups:
- MEC Cohort 1000 mg/Day (600mg AM, 400mg PM): Participants with advanced or recurrent mucoepidermoid carcinoma (MEC) who received PLX3397.
- PVNS Cohort 1000 mg/Day (600mg AM, 400mg PM): Participants with advanced pigmented villonodular synovitis (PVNS) who received PLX3397.
- GIST Cohort 1000 mg/Day (600mg AM, 400mg PM): Participants with advanced gastrointestinal stromal tumor (GIST) who received PLX3397.
- ATC Cohort 1000 mg/Day (600mg AM, 400mg PM): Participants with anaplastic thyroid carcinoma (ATC) who received PLX3397.
- Malignant Effusion Cohort 1000 mg/Day (600mg AM, 400mg PM): Participants with advanced solid tumors with malignant effusion who received PLX3397.
- Other Solid Tumor Type Cohort 1000 mg/Day (600mg AM, 400mg PM): Participants with other solid tumor types who received PLX3397.
Arm/Group | Dose Escalation Cohort 1: 200 mg QD | Dose Escalation Cohort 2: 300 mg QD | Dose Escalation Cohort 3: 400 mg QD | Dose Escalation Cohort 4: 600 mg QD | Dose Escalation Cohort 5: 900 mg/Day (500mg AM, 400mg PM) | Dose Escalation Cohort 6: 1200 mg/Day (600mg BID) | Dose Escalation Cohort 7: 1000 mg/Day (500mg BID) | MEC Cohort 1000 mg/Day (600mg AM, 400mg PM) | PVNS Cohort 1000 mg/Day (600mg AM, 400mg PM) | GIST Cohort 1000 mg/Day (600mg AM, 400mg PM) | ATC Cohort 1000 mg/Day (600mg AM, 400mg PM) | Malignant Effusion Cohort 1000 mg/Day (600mg AM, 400mg PM) | Other Solid Tumor Type Cohort 1000 mg/Day (600mg AM, 400mg PM)
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/6 | 1/6 | 0/6 | 0/7 | 1/6 | 0/7 | 1/4 | 0/39 | 3/11 | 1/9 | 1/8 | 1/20
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/6 | 0/6 | 0/6 | 1/7 | 1/6 | 3/7 | 2/4 | 5/39 | 4/11 | 1/9 | 2/8 | 3/20
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 6/6 | 6/6 | 6/7 | 6/6 | 7/7 | 4/4 | 39/39 | 11/11 | 8/9 | 8/8 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Cohort 1: 200 mg QD (N=3) | Dose Escalation Cohort 2: 300 mg QD (N=6) | Dose Escalation Cohort 3: 400 mg QD (N=6) | Dose Escalation Cohort 4: 600 mg QD (N=6) | Dose Escalation Cohort 5: 900 mg/Day (500mg AM, 400mg PM) (N=7) | Dose Escalation Cohort 6: 1200 mg/Day (600mg BID) (N=6) | Dose Escalation Cohort 7: 1000 mg/Day (500mg BID) (N=7) | MEC Cohort 1000 mg/Day (600mg AM, 400mg PM) (N=4) | PVNS Cohort 1000 mg/Day (600mg AM, 400mg PM) (N=39) | GIST Cohort 1000 mg/Day (600mg AM, 400mg PM) (N=11) | ATC Cohort 1000 mg/Day (600mg AM, 400mg PM) (N=9) | Malignant Effusion Cohort 1000 mg/Day (600mg AM, 400mg PM) (N=8) | Other Solid Tumor Type Cohort 1000 mg/Day (600mg AM, 400mg PM) (N=20)
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Cohort 1: 200 mg QD (N=3) | Dose Escalation Cohort 2: 300 mg QD (N=6) | Dose Escalation Cohort 3: 400 mg QD (N=6) | Dose Escalation Cohort 4: 600 mg QD (N=6) | Dose Escalation Cohort 5: 900 mg/Day (500mg AM, 400mg PM) (N=7) | Dose Escalation Cohort 6: 1200 mg/Day (600mg BID) (N=6) | Dose Escalation Cohort 7: 1000 mg/Day (500mg BID) (N=7) | MEC Cohort 1000 mg/Day (600mg AM, 400mg PM) (N=4) | PVNS Cohort 1000 mg/Day (600mg AM, 400mg PM) (N=39) | GIST Cohort 1000 mg/Day (600mg AM, 400mg PM) (N=11) | ATC Cohort 1000 mg/Day (600mg AM, 400mg PM) (N=9) | Malignant Effusion Cohort 1000 mg/Day (600mg AM, 400mg PM) (N=8) | Other Solid Tumor Type Cohort 1000 mg/Day (600mg AM, 400mg PM) (N=20)
Fatigue (General disorders) | 0 | 3 | 1 | 3 | 5 | 2 | 3 | 2 | 36 | 7 | 5 | 6 | 12
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 3 | 1 | 28 | 4 | 0 | 1 | 10
Nausea (Gastrointestinal disorders) | 1 | 3 | 3 | 4 | 4 | 2 | 2 | 1 | 26 | 4 | 3 | 5 | 9
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 1 | 4 | 2 | 3 | 4 | 0 | 9 | 3 | 5 | 4 | 9
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 15 | 2 | 1 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 0 | 2 | 2 | 2 | 16 | 4 | 2 | 3 | 2
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 15 | 1 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 3 | 2 | 3 | 3 | 1 | 3 | 1 | 14 | 1 | 3 | 2 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 14 | 0 | 0 | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 11 | 2 | 0 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 11 | 1 | 1 | 0 | 4
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 7 | 4 | 2 | 2 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 9 | 1 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 9 | 2 | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 4 | 3 | 2 | 3 | 2 | 0 | 10 | 3 | 0 | 2 | 6
Headache (Nervous system disorders) | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 13 | 1 | 0 | 0 | 5
Oedema peripheral (General disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 15 | 2 | 2 | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 1 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 6 | 0 | 2 | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 2
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 3 | 0 | 0 | 1 | 11 | 2 | 4 | 3 | 6
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 5 | 1 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 8 | 1 | 1 | 0 | 2
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 3 | 2 | 1 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 4 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 1
Retching (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 1 | 2 | 1 | 0 | 2 | 0 | 3 | 1 | 1 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 2 | 0 | 2 | 1 | 0 | 2 | 1 | 1 | 1 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Infusion site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 9 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 1 | 11 | 0 | 1 | 0 | 2
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 0 | 1 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 2 | 1 | 2 | 1 | 2 | 0 | 2 | 3 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 8 | 1 | 3 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 6 | 0 | 0 | 1 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 7 | 0 | 0 | 0 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 24 | 0 | 0 | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 5 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 11 | 0 | 1 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 0 | 0 | 0 | 4
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Occult blood positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 6 | 0 | 0 | 0 | 3
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 5 | 1 | 1 | 0 | 3
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 5 | 1 | 2 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 1 | 1 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Distractibility (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impulsive behaviour (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 5 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 6 | 0 | 0 | 0 | 2
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0
Lacrimation increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Myodesopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaphylactic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electromechanical dissociation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal septum ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sleep talking (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestine obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Superior vena caval occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Exophthalmos (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT01004861/Prot_SAP_001.pdf